CLINICAL TRIAL: NCT07150624
Title: Polyene Phosphatidylcholine Injection for the Treatment of Perioperative Liver Injury With Laparoscopic Hemihepatectomy in Hepatocellular Carcinoma: a Multicenter Randomized Controlled Study
Brief Title: The Treatment of Liver Injury After Liver Resection With Polyene Phosphatidylcholine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); The Second Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Bengbu Medical University (Other); First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXPJJH125002-2503
Record Dates: First submitted 2025-08-21; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC); Liver Diseases
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Experimental Group
- control group (Active Comparator)
  Interventions: Drug: control group

INTERVENTIONS:
Drug: Experimental Group — Receiving 930mg of polyene phosphatidylcholine injection one day before the operation,twice a day. And 930mg of polyene phosphatidylcholine injection,twice a day, combined with 100mg of magnesium isoglycyrrhizinate injection once a day，from the 1st to the 5th day after the operation.
  Arms: Experimental group
Drug: control group — Receiving 100mg of magnesium isoglycyrrhizinate injection once a day，from the 1st to the 5th day after the operation.
  Arms: control group

SUMMARY:
A multicenter, open-label, randomized, controlled study. It is proposed to evaluate the treatment plan of receiving 930mg polyene phosphatidylcholine injection one day before the operation, twice a day, and 930mg polyene phosphatidylcholine injection twice a day,combined with 100mg of magnesium isoglycyrrhizinate injection once a day,from the 1st to the 5th day after the operation. Compared with the monotherapy regimen of no liver protection treatment before the operation and receiving magnesium isoglycyrrhizinate injection 100mg once a day from the 1st to the 5th day after the operation.The efficacy and safety of treating postoperative liver function injury in patients undergoing laparoscopic hemihepatectomy for hepatocellular carcinoma were compared.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as HCC through imaging and laboratory tests, and capable of undergoing laparoscopic anatomical resection
2. Those who plan to undergo right or left hemi-liver resection
3. During the operation, the Pringle method was used to block the first hepatic portal. Each block lasted for no more than 15 minutes, and the blocking procedure was performed 2 to 4 times.
4. Age: 18 - 70 years old. Gender: Open to both male and female. Body Mass Index (BMI): 18.5 - 28 kg/m2
5. Child-Pugh grade A or B, with a score of ≤ 7; ASA grades I to III
6. Preoperative ICG R15 was less than 10%, and the residual liver volume was more than 40% of the standard liver volume
7. A single HCC (hepatocellular carcinoma), with a tumor diameter less than 10 cm, without distant metastasis or invasion of the portal vein system
8. Preoperative ALT was less than 2 times the upper limit of normal
9. Before being enrolled in the study, the patient had no history of any other treatments, such as portal vein embolization, TACE or systemic anti-tumor drug therapy.
10. No liver-damaging treatment drugs were used within two weeks prior to enrollment.

Exclusion Criteria:

1. Reserve liver vascular damage, including: reconstruction after severance, ligation, embolization, thrombosis, etc
2. Combined with abnormal coagulation function (prothrombin time prolonged by more than 3 seconds)
3. Combining obstructive jaundice, severe heart disease, severe kidney disease and other serious illnesses
4. During the operation, microwave treatment or a combination of microwave treatment was adopted
5. More than 4 times of blocking at the first hepatic hilum, or a single blocking duration longer than 15 minutes
6. Non-anatomic liver resection, where the remaining liver contains large areas of ischemic/edematous regions
7. More than 1000ml of blood transfusion during the operation
8. During the operation, an extra-hepatic disease was discovered. Other organs except the gallbladder needed to be removed simultaneously
9. During the operation, other intrahepatic lesions were discovered, which required combination with other surgeries, such as ablation or choledochojejunostomy
10. Diseases that have previously received systemic treatment with glucocorticoids, such as chronic kidney disease, inflammatory diseases, or other immune system-related disorders
11. Psychosis, severe neurosis, those who cannot cooperate with this experiment
12. Participated in other clinical trials within the previous 3 months before enrollment
13. Allergy or intolerance to benzoic acid, or to the study drug
14. Pregnant and lactating women
15. The researchers believe that any participants who have any other factors that would make them unsuitable for this trial should not be included

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The average change of ALT on the 5th day after the operation | The 5th day after the operation

SECONDARY OUTCOMES:
The average change of ALT on the 1th day after the operation | The 1th day after the operation
The average change of ALT on the 3th day after the operation | The 3th day after the operation
The rate of ALT returning to normal on the 5th day after the operation | The 5th day after the operation
The rate of AST returning to normal on the 5th day after the operation | The 5th day after the operation
AEs | Observation period 5 days after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No